CLINICAL TRIAL: NCT02314000
Title: WHISPER - A Randomized Controlled Study to Evaluate the Effectiveness of the Precision Spinal Cord Stimulator System at Sub-Perception Amplitude
Brief Title: Effectiveness of the Precision Spinal Cord Stimulator System at Sub-Perception Amplitude
Acronym: WHISPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A4046; 90987574 (Other: Boston Scientific (study protocol number))
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Results first posted 2019-04-12 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SCS starting with supra-perception (Active Comparator): Precision or Precision Spectra Spinal Cord Stimulator System programmed at supra-perception followed by sub-perception SCS
  Interventions: Device: Precision or Precision Spectra Spinal Cord Stimulator System
- SCS starting with sub-perception amplitude (Experimental): Precision or Precision Spectra Spinal Cord Stimulator System programmed at sub-perception followed by supra-perception SCS
  Interventions: Device: Precision or Precision Spectra Spinal Cord Stimulator System

INTERVENTIONS:
Device: Precision or Precision Spectra Spinal Cord Stimulator System

SUMMARY:
To demonstrate sustained clinically significant pain relief in patients with chronic pain when using the Boston Scientific Precision Spinal Cord Stimulator (SCS) System at sub-perception amplitude

DETAILED DESCRIPTION:
To demonstrate sustained clinically significant pain relief in patients when using the Boston Scientific Precision Spinal Cord Stimulator (SCS) System at sub-perception amplitude

ELIGIBILITY:
Key Inclusion Criteria:

1. Complaint of chronic pain of the trunk and/or limbs
2. Willing and able to comply with all protocol-required procedures and assessments/evaluations; able to independently read and complete all questionnaires and assessments provided in English
3. Subject signed a valid, Institutional Review Board (IRB)-approved informed consent form (ICF) provided in English

Key Exclusion Criteria:

1. Meets any contraindication in the Precision SCS system per locally applicable Directions for Use (DFU)
2. Any pain-related diagnosis or medical/psychological condition that, in the clinician's best judgment, might confound reporting of study outcomes

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roshini Jain, M.S., Study Director — Boston Scientific Neuromodulation Corporation
Locations (26):
- United States (26):
  - MORE Foundation, Phoenix, Arizona
  - Coastal Pain & Spinal Diagnostics, Carlsbad, California
  - Kaiser Foundation Hospital - Redwood City, Redwood City, California
  - University of California, Davis Medical Center, Sacramento, California
  - Clearwater Pain Management, Clearwater, Florida
  - Tallahassee Neurological Clinic, PA, Tallahassee, Florida
  - Shepherd Center, Atlanta, Georgia
  - Orthopedic Research Foundation, Savannah, Georgia
  - American Health Network of Indiana, LLC, Muncie, Indiana
  - Forest Health Medical Center, Ypsilanti, Michigan
  - Jackson Anesthesia Pain Center, LLC, Jackson, Mississippi
  - Comprehensive Pain & Rehabilitation, Pascagoula, Mississippi
  - KC Pain Centers, Lee's Summit, Missouri
  - Mercy Medical Research Institute, Springfield, Missouri
  - Vidant Roanoke - Chowan Hospital Pain Center, Ahoskie, North Carolina
  - The Center for Clinical Research, LLC, Winston-Salem, North Carolina
  - University of Cincinnati Physicians Company, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Western Reserve Hospital, Cuyahoga Falls, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Florence Neurosurgery and Spine, Florence, South Carolina
  - PCPMG Clinical Research Unit, LLC, Greenville, South Carolina
  - TBI Clinical Research, L.L.C., Plano, Texas
  - Swedish Medical Center, Seattle, Washington

REFERENCES:
- [Derived] North J, Loudermilk E, Lee A, Sachdeva H, Kaiafas D, Washabaugh E, Sheth S, Scowcroft J, Mekhail N, Lampert B, Yearwood T, Shaw E, Atallah J, McLeod C, Han J, Yu C, Sedrak M, Lucas R, Trobridge A, Hegarty J, Miller N, Chen L, Jain R. Outcomes of a Multicenter, Prospective, Crossover, Randomized Controlled Trial Evaluating Subperception Spinal Cord Stimulation at </=1.2 kHz in Previously Implanted Subjects. Neuromodulation. 2020 Jan;23(1):102-108. doi: 10.1111/ner.13015. Epub 2019 Jul 2. PMID 31265205

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolled subjects underwent study eligibility to determine if they can continue in the study. Following completion of study eligibility, subjects were randomized to the cross-over phase.
Groups:
- SCS Starting With Supra-perception Amplitude: Precision or Precision Spectra Spinal Cord Stimulator System programmed starting with supra-perception followed by sub-perception amplitude.
  Precision or Precision Spectra Spinal Cord Stimulator System
- SCS Starting With Sub-perception Amplitude: Precision or Precision Spectra Spinal Cord Stimulator System programmed starting with sub-perception and followed by supra-perception amplitude.
  Precision or Precision Spectra Spinal Cord Stimulator System
Period: Overall Study
Arm/Group | SCS Starting With Supra-perception Amplitude | SCS Starting With Sub-perception Amplitude
Started | 75 | 65
Completed | 62 | 57
Not Completed | 13 | 8

BASELINE CHARACTERISTICS:
Groups:
- SCS Starting at Supra-perception Amplitude: Precision or Precision Spectra Spinal Cord Stimulator System programmed starting at supra-perception and followed by sub-perception amplitude.
  Precision or Precision Spectra Spinal Cord Stimulator System
- SCS Starting at Sub-perception Amplitude: Precision or Precision Spectra Spinal Cord Stimulator System starting at sub-perception and followed by supra-perception amplitude.
  Precision or Precision Spectra Spinal Cord Stimulator System
- Total: Total of all reporting groups
Arm/Group | SCS Starting at Supra-perception Amplitude | SCS Starting at Sub-perception Amplitude | Total
Number analyzed (Participants) | 75 | 65 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (11.9) | 58.8 (10.7) | 59.8 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 39 | 83
  Male | 31 | 26 | 57

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With 50% or Greater Reduction in Overall Pain Intensity From Baseline
Description: Proportion of subjects with 50% or greater reduction in overall pain intensity from baseline with supra and sub perception amplitude with no increase in average daily medication intake to treat pain
Time Frame: 90 days post activation
Population: Due to the nature of crossover study design, all subjects contributed towards each arm, as reflected in the number of participants.
Measure: Count of Participants; unit: Participants
Groups:
- SCS With Supra-perception Amplitude: Precision or Precision Spectra Spinal Cord Stimulator System programmed at supra-perception amplitude
  Precision or Precision Spectra Spinal Cord Stimulator System
- SCS With Sub-perception Amplitude: Precision or Precision Spectra Spinal Cord Stimulator System programmed at sub-perception amplitude
  Precision or Precision Spectra Spinal Cord Stimulator System
Arm/Group | SCS With Supra-perception Amplitude | SCS With Sub-perception Amplitude
Number analyzed (Participants) | 119 | 118
Participants | 32 | 41

ADVERSE EVENTS:
Time Frame: Adverse events up to end of cross over period - approximately upto 180 days after randomization
Description: Adverse events up to end of cross over period - approximately upto 180 days after randomization
Groups:
- All Study Patients Through End of Randomized Phase: All adverse events reported through end of randomized phase
- SCS With Supra Perception Amplitude; SCS With Subperception Amplitude: All adverse events during SCS with supra perception amplitude
Arm/Group | All Study Patients Through End of Randomized Phase | SCS With Supra Perception Amplitude | SCS With Subperception Amplitude
All-Cause Mortality (participants affected / at risk) | 0/140 | 0/140 | 0/140
Serious Adverse Events (participants affected / at risk) | 7/140 | 3/140 | 4/140
Other Adverse Events (participants affected / at risk) | 0/140 | 0/140 | 0/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Patients Through End of Randomized Phase (N=140) | SCS With Supra Perception Amplitude (N=140) | SCS With Subperception Amplitude (N=140)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Diverticular Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Enterocolitis Heamorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Post Procedure Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical study agreement that restricts PI until official study manuscript is available.